CLINICAL TRIAL: NCT02853305
Title: A Phase III Randomized, Controlled Clinical Trial of Pembrolizumab With or Without Platinum-Based Combination Chemotherapy Versus Chemotherapy in Subjects With Advanced or Metastatic Urothelial Carcinoma
Brief Title: Study of Pembrolizumab With or Without Platinum-based Combination Chemotherapy Versus Chemotherapy Alone in Urothelial Carcinoma (MK-3475-361/KEYNOTE-361)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3475-361; 163458 (Registry Identifier: JAPIC-CTI); MK-3475-361 (Other: Merck Protocol Number); 2015-005731-41 (EudraCT Number)
Record Dates: First submitted 2016-07-29; First posted 2016-08-02 (Estimated); Results first posted 2021-05-20 (Actual); Last update posted 2023-09-08 (Actual); Status verified 2023-08

CONDITIONS: Urothelial Carcinoma Associated 1 RNA, Human
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL2, PD-L2)
MeSH Terms: conditions — Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Cisplatin; Carboplatin; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab + ST Chemotherapy (Pembro Combo) (Experimental): Participants receive pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for a maximum of 35 doses PLUS standard therapy (ST) chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle + gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle, OR carboplatin at an area under the curve 5 (AUC 5) (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle + gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle. Eligible participants who stop pembrolizumab with Stable Disease (SD) or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab; Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine
- Pembrolizumab (Pembro) (Experimental): Participants receive pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for a maximum of 35 doses. Eligible participants who stop pembrolizumab with SD or better but progress after discontinuation may be able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
  Interventions: Biological: Pembrolizumab
- ST Chemotherapy (Chemo) (Active Comparator): Participants receive ST chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle + gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle OR carboplatin at AUC 5 (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle + gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle.
  Interventions: Drug: Cisplatin; Drug: Carboplatin; Drug: Gemcitabine

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab (Pembro); Pembrolizumab + ST Chemotherapy (Pembro Combo)
Drug: Cisplatin — IV infusion
  Arms: Pembrolizumab + ST Chemotherapy (Pembro Combo); ST Chemotherapy (Chemo)
Drug: Carboplatin — IV infusion
  Arms: Pembrolizumab + ST Chemotherapy (Pembro Combo); ST Chemotherapy (Chemo)
Drug: Gemcitabine — IV infusion
  Arms: Pembrolizumab + ST Chemotherapy (Pembro Combo); ST Chemotherapy (Chemo)

SUMMARY:
The purpose of this study is to determine the efficacy and safety of pembrolizumab (pembro, MK-3475) with or without chemotherapy versus chemotherapy alone in participants with advanced or metastatic urothelial carcinoma (bladder cancer).

The primary hypotheses are that pembrolizumab plus chemotherapy is superior to chemotherapy alone with respect to Progression-free Survival (PFS) and Overall Survival (OS) in all participants, and that pembrolizumab alone is superior to chemotherapy alone with respect to OS in all participants and in participants with programmed cell death ligand 1 (PD-L1) positive tumors (Combined Positive Score [CPS] ≥10%).

DETAILED DESCRIPTION:
As specified by the protocol, the study hypotheses will be evaluated by comparing the pembro combo arm or pembro arm separately to the chemo arm.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of advanced/unresectable (inoperable) or metastatic urothelial carcinoma of the renal pelvis, ureter [upper urinary tract], bladder, or urethra. Both transitional cell and mixed transitional/non- transitional cell histologies are allowed, but transitional cell carcinoma must be the predominant histology.
* Has measurable disease based on RECIST 1.1 as determined by the local site investigator/radiology assessment.
* Has received no prior systemic chemotherapy for advanced or metastatic urothelial carcinoma, with the following exceptions:

  * Neoadjuvant platinum-based chemotherapy with recurrence >12 months from completion of therapy is permitted.
  * Adjuvant platinum-based chemotherapy following radical cystectomy with recurrence >12 months from completion of therapy is permitted.
* Has provided tissue for biomarker analysis from an archival tissue sample or newly obtained core or excisional biopsy of a tumor lesion not previously irradiated from a muscle invasive urothelial carcinoma or a metastatic biopsy, originally from the original tumor.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2.
* Demonstrates adequate organ function.
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of pembrolizumab or 180 days after chemotherapy treatment.
* Male participants of childbearing potential must agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of pembrolizumab or 180 days after chemotherapy treatment.

Exclusion Criteria:

* Has disease that is suitable for local therapy administered with curative intent.
* Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigation device within 4 weeks of the first dose of study drug.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to randomization.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has had a prior anti-cancer monoclonal antibody (mAb) for direct anti-neoplastic treatment within 4 weeks prior to the first dose of study drug (6 weeks for nitrosoureas or mitomycin C) or who has not recovered (i.e., ≤ Grade 1 or at Baseline) from adverse events (AEs) due to mAbs administered more than 4 weeks earlier.
* Has not recovered (i.e., AE ≤ Grade 1 or at Baseline) from AEs due to a previously administered agent.
* Has a known additional malignancy that is progressing or requires active treatment within the past 5 years.

  * Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
  * A history of prostate cancer that was identified incidentally following cystoprostatectomy for bladder cancer is acceptable, provided that the following criteria are met: Stage T2N0M0 or lower; Gleason score ≤6; Prostate-specific Antigen (PSA) level undetectable.
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a known history of active tuberculosis (TB).
* Has an active infection requiring systemic therapy.
* Has a history of severe hypersensitivity reaction (e.g. generalized rash/erythema, hypotension, bronchospasm, angioedema or anaphylaxis) to pembrolizumab, gemcitabine, carboplatin, or cisplatin or their analogs and/or to any of their excipients.
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial. Is a known regular user (including "recreational use") of any illicit drug(s) or had a recent history (within the last year) of drug or alcohol abuse.
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of pembrolizumab or 180 days after the last dose of chemotherapy treatment.
* Has received prior therapy with an anti-PD-1, or anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137).
* Has a known history of human immunodeficiency virus (HIV).
* Has known active hepatitis B or hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1010 (Actual)
Dates: Start 2016-09-15 (Actual); Primary Completion 2020-04-29 (Actual); Study Completion 2022-09-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Giannatempo P, Machiels JP, Sassa N, Arranz JA, Fujii Y, Su WP, Keam B, Culine S, Shen YC, Langa JM, Sarid D, Aarts M, Calabro F, Rosenbaum E, Moreno BH, Bavle A, Xu JZ, Rha SY. Impact of Histology on Clinical Outcomes of Pembrolizumab Monotherapy in Patients With Advanced or Metastatic Urothelial Carcinoma in the Phase 3 KEYNOTE-045 and KEYNOTE-361 Trials. Clin Genitourin Cancer. 2025 Apr;23(2):102273. doi: 10.1016/j.clgc.2024.102273. Epub 2024 Nov 15. PMID 40037029
- [Derived] Powles T, Chang YH, Yamamoto Y, Munoz J, Reyes-Cosmelli F, Peer A, Cohen G, Yu EY, Lorch A, Bavle A, Homet Moreno B, Markensohn J, Edmondson M, Chen C, Cristescu R, Pena C, Lunceford J, Gunduz S. Pembrolizumab for advanced urothelial carcinoma: exploratory ctDNA biomarker analyses of the KEYNOTE-361 phase 3 trial. Nat Med. 2024 Sep;30(9):2508-2516. doi: 10.1038/s41591-024-03091-7. Epub 2024 Jun 1. PMID 38823511
- [Derived] Topp BG, Channavazzala M, Mayawala K, De Alwis DP, Rubin E, Snyder A, Wolchok JD, Ribas A. Tumor dynamics in patients with solid tumors treated with pembrolizumab beyond disease progression. Cancer Cell. 2023 Sep 11;41(9):1680-1688.e2. doi: 10.1016/j.ccell.2023.08.004. PMID 37699333
- [Derived] Powles T, Csoszi T, Ozguroglu M, Matsubara N, Geczi L, Cheng SY, Fradet Y, Oudard S, Vulsteke C, Morales Barrera R, Flechon A, Gunduz S, Loriot Y, Rodriguez-Vida A, Mamtani R, Yu EY, Nam K, Imai K, Homet Moreno B, Alva A; KEYNOTE-361 Investigators. Pembrolizumab alone or combined with chemotherapy versus chemotherapy as first-line therapy for advanced urothelial carcinoma (KEYNOTE-361): a randomised, open-label, phase 3 trial. Lancet Oncol. 2021 Jul;22(7):931-945. doi: 10.1016/S1470-2045(21)00152-2. Epub 2021 May 26. PMID 34051178
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with advanced or metastatic urothelial carcinoma were recruited to examine the efficacy and safety of pembrolizumab plus chemotherapy (pembro combo) versus pembrolizumab alone (pembro) or chemotherapy alone (chemo).
Pre-assignment Details: 1,010 participants were randomized 1:1:1 to receive pembrolizumab plus chemotherapy, pembrolizumab alone, or chemotherapy alone. Per protocol, response/progression or adverse events (AEs) that occurred during the second course were not counted towards efficacy outcome measures or safety outcome measures, respectively.
Groups:
- Pembrolizumab + ST Chemotherapy (Pembro Combo): Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for a maximum of 35 doses PLUS standard therapy (ST) chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle + gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle, OR carboplatin at an area under the curve 5 (AUC 5) (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle + gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle. Eligible participants who stopped pembrolizumab with Stable Disease (SD) or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- Pembrolizumab (Pembro): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for a maximum of 35 doses. Eligible participants who stopped pembrolizumab with SD or better but progressed after discontinuation may have been able to initiate a second course of pembrolizumab for up to 17 cycles (up to approximately 1 additional year) at the investigator's discretion.
- ST Chemotherapy (Chemo): Participants received ST chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle OR carboplatin at AUC 5 (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle.
Period: Overall Study
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Started | 351 | 307 | 352
Received First Course of Pembrolizumab | 349 (Includes 2 participants randomized to Pembrolizumab alone) | 302 | 342
Received Second Course of Pembrolizumab | 14 | 15 | 0
Completed | 0 | 0 | 0
Not Completed | 351 | 307 | 352
Not completed — Death | 287 | 249 | 300
Not completed — Withdrawal by Subject | 2 | 8 | 3
Not completed — Transferred to Extension Study | 46 | 30 | 25
Not completed — Did Not Continue on Extension Study | 16 | 20 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo) | Total
Number analyzed (Participants) | 351 | 307 | 352 | 1010
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.3 (9.2) | 67.0 (10.1) | 68.0 (9.6) | 67.8 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 79 | 79 | 90 | 248
  Male | 272 | 228 | 262 | 762
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 25 | 32 | 83
  Not Hispanic or Latino | 269 | 231 | 261 | 761
  Unknown or Not Reported | 56 | 51 | 59 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 64 | 47 | 70 | 181
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 4 | 8
  White | 243 | 212 | 235 | 690
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 42 | 42 | 42 | 126
PD-L1 CPS Status-IVRS [Count of Participants; unit: Participants] — The Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) Status indicates tumor PD-L1 positivity using both tumor cells and inflammatory cells that are positive for PD-L1 by immunohistochemistry (IHC). Higher percentages of PD-L1 CPS staining corresponded to higher positivity of PD-L1 on a tumor. The number of participants with CPS <10% and CPS ≥10% at baseline randomization by Interactive Voice Response System (IVRS) is presented
  Participants
    PD-L1 CPS<10 | 192 | 148 | 193 | 533
    PD-L1 CPS≥10 | 159 | 159 | 159 | 477
Investigator Choice of Cisplatin or Carboplatin - IVRS [Count of Participants; unit: Participants] — The Investigator's choice of chemotherapy drug (cisplatin or carboplatin) at baseline randomization by IVRS is presented.
  Participants
    Cisplatin | 160 | 138 | 160 | 458
    Carboplatin | 191 | 169 | 192 | 552

OUTCOME MEASURES:

1. Primary Outcome: Pembro Combo vs Chemo: Progression-free Survival (PFS) Using Response Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: PFS was defined as the time from randomization to the first documented progressive disease (PD) per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study.
  Per protocol, PFS in the pembro combo arm was compared to the chemo arm as a pre-specified primary analysis of the Intent-To-Treat (ITT) population (all randomized participants). PFS is reported here for all participants in the pembro combo arm and chemo arm. Per protocol, PFS was compared separately between all participants of the pembro arm and chemo arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: All participants in the ITT population randomized to the pembro combo arm and chemo arm were included in the analysis. Per protocol, the pembro arm was compared to the chemo arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab + ST Chemotherapy (Pembro Combo): Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle for a maximum of 35 doses PLUS standard therapy (ST) chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle, OR carboplatin at an area under the curve 5 (AUC 5) (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle.
- Pembrolizumab (Pembro): Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle for a maximum of 35 doses.
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 0 | 352
Months | 8.3 [7.5 to 8.5] |  | 7.1 [6.4 to 7.9]
Statistical Analysis 1: Comparison: Pembrolizumab + ST Chemotherapy (Pembro Combo) vs ST Chemotherapy (Chemo); PFS in all participants of the pembro combo arm was compared to PFS in all participants of the chemo arm to address the first primary hypothesis (superiority to chemo). The hazard ratio (HR) and its 95% confidence interval (CI) were estimated using a stratified Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Superiority; p = 0.0033, Stratified Log-Rank; The treatment difference in PFS was assessed by the stratified log-rank test; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.65 to 0.93]

2. Primary Outcome: Pembro Combo vs Chemo: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro combo arm was compared to the chemo arm as a pre-specified primary analysis of the ITT population (all randomized participants). OS is reported here for all participants in the pembro combo arm and chemo arm. Per protocol, OS was compared separately between all participants of the pembro arm and chemo arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 0 | 352
Months | 17.0 [14.5 to 19.5] |  | 14.3 [12.3 to 16.7]
Statistical Analysis 1: Comparison: Pembrolizumab + ST Chemotherapy (Pembro Combo) vs ST Chemotherapy (Chemo); OS in all participants of the pembro combo arm was compared to OS in all participants of the chemo arm to address the second primary hypothesis (superiority to chemo). The HR and its 95% CI were estimated using a stratified Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Superiority; p = 0.0407, Stratified Log-Rank; The treatment difference in OS was assessed by the stratified log-rank test; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.72 to 1.02]

3. Primary Outcome: Pembro vs Chemo: OS in Participants With Programmed Cell Death Ligand 1 (PD-L1) Combined Positive Score (CPS) ≥10%
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the CPS ≥10% subset of the pembro arm was compared to OS in the CPS ≥10% subset of the chemo arm for this endpoint as a pre-specified primary analysis of the ITT population. OS is reported here for all participants in the pembro arm and chemo arm who were PD-L1 CPS ≥10%. Per protocol, OS in the CPS ≥10% subset of the pembro combo arm was not a pre-specified analysis of the ITT population and is not presented.
Time Frame: Up to approximately 42 months
Population: All participants in the ITT population randomized to the pembro arm and chemo arm who were PD-L1 CPS ≥10% were included in the analysis. Per protocol, the pembro combo arm was not pre-specified as part of this analysis and is not included.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 160 | 158
Months |  | 16.1 [13.6 to 19.9] | 15.2 [11.6 to 23.3]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); OS in CPS≥10 participants of the pembro arm was compared to OS in CPS≥10 participants of the chemo arm. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) at baseline; Test type: Other; No formal hypothesis testing was performed; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.77 to 1.32]

4. Primary Outcome: Pembro vs Chemo: OS
Description: OS was defined as the time from randomization to death due to any cause. Participants without documented death at the time of the final analysis were censored at the date of the last follow-up. Per protocol, OS in the pembro arm was compared to the chemo arm as a pre-specified primary analysis of the ITT population (all randomized participants). OS is reported here for all participants in the pembro arm and chemo arm. Per protocol, OS was compared separately between all participants of the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: All participants in the ITT population randomized to the pembro arm and chemo arm were included in the analysis. Per protocol, the pembro combo arm was compared to the chemo arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 307 | 352
Months |  | 15.6 [12.1 to 17.9] | 14.3 [12.3 to 16.7]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); OS in all participants of the pembro arm was compared to OS in all participants of the chemo arm. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.77 to 1.11]

5. Secondary Outcome: Pembro vs Chemo: PFS Using RECIST 1.1 as Assessed by BICR
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study.
  Per protocol, PFS in the pembro arm was compared to the chemo arm as a pre-specified analysis of the ITT population (all randomized participants). PFS is reported here for all participants in the pembro arm and chemo arm. Per protocol, PFS was compared separately between all participants of the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 307 | 352
Months |  | 3.9 [2.3 to 5.1] | 7.1 [6.4 to 7.9]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); PFS in all participants of the pembro arm was compared to PFS in all participants of the chemo arm. The comparison was based on a Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Hazard Ratio (HR) = 1.32, 95% CI 2-sided [1.09 to 1.58]

6. Secondary Outcome: Number of Participants Who Experience an Adverse Event (AE)
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that experienced at least one AE was reported for each treatment arm.
Time Frame: Up to approximately 55 months
Population: All randomized participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 349 | 302 | 342
Participants | 348 | 289 | 341

7. Secondary Outcome: Number of Participants Who Discontinue Study Drug Due to an AE
Description: An AE was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have to have a causal relationship with this treatment. An AE could therefore be any unfavourable and unintended sign, symptom, or disease temporally associated with the use of a medicinal product or protocol-specified procedure, whether or not considered related to the medicinal product or protocol-specified procedure. Any worsening of a pre-existing condition that was temporally associated with the use of the Sponsor's product was also an AE. The number of participants that discontinued any study drug due to an AE was reported for each treatment arm.
Time Frame: Up to approximately 52 months
Population: All randomized participants who received at least 1 dose of trial treatment were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 349 | 302 | 342
Participants | 108 | 48 | 62

8. Secondary Outcome: Pembro Combo vs Chemo: Objective Response Rate (ORR) Using RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants in the analysis population who had a Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: ≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, ORR in the pembro combo arm was compared to the chemo arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR for all participants in the pembro combo arm and chemo arm. Per protocol, ORR was compared separately between participants of the pembro arm and chemo arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 0 | 352
Percentage of Participants | 54.7 [49.3 to 60.0] |  | 44.9 [39.6 to 50.2]
Statistical Analysis 1: Comparison: Pembrolizumab + ST Chemotherapy (Pembro Combo) vs ST Chemotherapy (Chemo); ORR in participants of the pembro combo arm was compared to ORR in participants of the chemo arm. The comparison was based on the Miettinen & Nurminen method stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Difference in Percentage = 9.8, 95% CI 2-sided [2.4 to 17.1]

9. Secondary Outcome: Pembro Combo vs Chemo: Duration of Response (DOR) Using RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based upon BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. DOR is reported here for all participants in the pembro combo arm and chemo arm who had CR or PR. Per protocol, DOR was assessed separately in responders of the pembro arm and chemo arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: All participants in the ITT population randomized to the pembro combo arm and chemo arm and who demonstrated a confirmed CR or PR were included in the analysis. Per protocol, the pembro arm was compared to the chemo arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 192 | 0 | 158
Months | 8.5 [8.2 to 11.4] |  | 6.2 [5.8 to 6.6]

10. Secondary Outcome: Pembro Combo vs Chemo: Disease Control Rate (DCR) Using RECIST 1.1 as Assessed by BICR
Description: DCR was defined as the percentage of participants who had a confirmed CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions), or Stable Disease (SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD]). Per protocol, DCR in the pembro combo arm was compared to the chemo arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced a confirmed CR, PR, or SD according to RECIST 1.1 as assessed by BICR was reported as the DCR for all participants in the pembro combo arm and chemo arm. Per protocol, DCR was compared separately between participants of the pembro arm and chemo arm and is presented later in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 0 | 352
Percentage of Participants | 80.3 [75.8 to 84.4] |  | 75.9 [71.0 to 80.2]
Statistical Analysis 1: Comparison: Pembrolizumab + ST Chemotherapy (Pembro Combo) vs ST Chemotherapy (Chemo); DCR in participants of the pembro combo arm was compared to DCR in participants of the chemo arm based on the Miettinen & Nurminen method stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Difference in Percentage = 4.5, 95% CI 2-sided [-1.6 to 10.6]

11. Secondary Outcome: Pembro vs Chemo: ORR Using RECIST 1.1 as Assessed by BICR
Description: ORR was defined as the percentage of participants in the analysis population who had a CR (disappearance of all target lesions) or a PR (≥30% decrease in the sum of diameters of target lesions) per RECIST 1.1. based upon BICR. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, ORR in the pembro arm was compared to the chemo arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced CR or PR is reported here as the ORR for all participants in the pembro arm and chemo arm. Per protocol, ORR was compared separately between participants of the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 307 | 352
Percentage of Participants |  | 30.3 [25.2 to 35.8] | 44.9 [39.6 to 50.2]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); ORR in participants of the pembro arm was compared to ORR in participants of the chemo arm. The comparison was based on the Miettinen & Nurminen method stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Superiority; No formal hypothesis testing was performed; Difference in Percentage = -14.8, 95% CI 2-sided [-22.0 to -7.4]

12. Secondary Outcome: Pembro vs Chemo: DOR Using RECIST 1.1 as Assessed by BICR
Description: For participants who demonstrated a confirmed CR (disappearance of all target lesions) or PR (at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 based upon BICR, DOR was defined as the time from first documented evidence of confirmed CR or PR until PD or death, whichever occurred first. DOR for participants who had not progressed or died at the time of analysis was censored at the date of their last tumor assessment. Per RECIST 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. DOR is reported here for all participants in the pembro arm and chemo arm who had CR or PR. Per protocol, DOR was assessed separately in responders of the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: All participants in the ITT population randomized to the pembro arm and chemo arm who demonstrated a confirmed CR or PR were included in the analysis. Per protocol, the pembro combo arm was compared to the chemo arm separately and not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 93 | 158
Months |  | 28.2 [13.5 to NA] — NA= DOR upper 95% confidence limit undefined because the DOR rate was not low enough at the time of the cut-off date | 6.2 [5.8 to 6.6]

13. Secondary Outcome: Pembro vs Chemo: DCR Using RECIST 1.1 as Assessed by BICR
Description: DCR was defined as the percentage of participants who had a CR (disappearance of all target lesions), PR (at least a 30% decrease in the sum of diameters of target lesions), or SD (neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD [at least a 20% increase in the sum of diameters of target lesions and an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD]). Per protocol, DCR in the pembro arm was compared to the chemo arm as a pre-specified secondary analysis of the ITT population. The percentage of participants who experienced a confirmed CR, PR, or SD according to RECIST 1.1 as assessed by BICR was reported as the DCR for all participants in the pembro arm and chemo arm. Per protocol, DCR was compared separately between participants of the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Up to approximately 42 months
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 307 | 352
Percentage of Participants |  | 47.2 [41.5 to 53.0] | 75.9 [71.0 to 80.2]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); DCR in participants of the pembro arm was compared to DCR in participants of the chemo arm based on the Miettinen & Nurminen method stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Difference in Percentage = -28.9, 95% CI 2-sided [-35.9 to -21.6]

14. Secondary Outcome: PFS Using RECIST 1.1 as Assessed by BICR at 6 Months
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, PFS was compared between arms as a pre-specified secondary analysis of the ITT population (all randomized participants). PFS is reported here for all participants at 6 months based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: 6 months
Population: All participants in the ITT population (all randomized) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 307 | 352
Percentage of Participants | 73.7 [68.6 to 78.0] | 43.6 [37.9 to 49.1] | 70.3 [64.8 to 75.0]

15. Secondary Outcome: PFS Using RECIST 1.1 as Assessed by BICR at 12 Months
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, PFS was compared between arms as a pre-specified secondary analysis of the ITT population (all randomized participants). PFS is reported here for all participants at 12 months based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: 12 months
Population: All participants in the ITT population (all randomized) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 307 | 352
Percentage of Participants | 33.7 [28.6 to 38.9] | 26.6 [21.6 to 31.9] | 20.9 [16.0 to 26.1]

16. Secondary Outcome: PFS Using RECIST 1.1 as Assessed by BICR at 18 Months
Description: PFS was defined as the time from randomization to the first documented PD per RECIST 1.1 based on BICR, or death due to any cause, whichever occurred first. Per RECIST 1.1, PD was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum had to demonstrate an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered PD. The sponsor allowed a maximum of 10 target lesions in total and 5 per organ on this study. Per protocol, PFS was compared between arms as a pre-specified secondary analysis of the ITT population (all randomized participants). PFS is reported here for all participants at 18 months based on the product-limit (Kaplan-Meier) method for censored data.
Time Frame: 18 months
Population: All participants in the ITT population (all randomized) were analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 351 | 307 | 352
Percentage of Participants | 23.0 [18.4 to 27.8] | 19.1 [14.7 to 24.0] | 13.5 [9.3 to 18.4]

17. Secondary Outcome: Pembro Combo vs Chemo: Change From Baseline to Week 18 in the European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Global Health Status/Quality of Life (Items 29 and 30) Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared between all participants of the pembro combo arm and the chemo arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared separately between all participants of the pembro arm and chemo arm and is presented later in the record.
Time Frame: Baseline, Week 18
Population: All participants in the ITT population randomized to the pembro combo arm and chemo arm who received at least 1 dose of study drug and who completed at least 1 EORTC-QLQ-C30 assessment were included in the analysis. Per protocol, the pembro arm was compared to the chemo arm separately and is not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 336 | 0 | 337
Score on a Scale | 2.54 [-0.08 to 5.16] |  | -0.14 [-2.91 to 2.63]
Statistical Analysis 1: Comparison: Pembrolizumab + ST Chemotherapy (Pembro Combo) vs ST Chemotherapy (Chemo); Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between all participants of the pembro combo arm and the chemo arm. Comparison based on constrained longitudinal data analysis (cLDA) model with GHS/QoL score as response variable, and with treatment by study visit interactions and stratification factors (investigator's choice of chemotherapy [cisplatin or carboplatin] and PD-L1 status [CPS<10 vs. CPS≥10]) at baseline as covariates; Test type: Other; No formal hypothesis testing was performed; Difference in LS Means = 2.68, 95% CI 2-sided [-0.76 to 6.12]

18. Secondary Outcome: Pembro Combo vs Chemo: Time to Deterioration (TTD) in the EORTC-QLQ-C30 GHS/QoL (Items 29 and 30) Combined Score
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD in GHS/QoL was defined as the time from first dose date to the first onset of a ≥10 point decrease from baseline in GHS/QoL combined score without confirmation. Per protocol, TTD in GHS/QoL combined score was compared between the pembro combo arm and chemo arm. TTD in GHS/QoL combined score was compared separately between the pembro arm and chemo arm and is presented later in the record.
Time Frame: Baseline up to approximately 25 months
Population: All participants in the ITT population randomized to the pembro combo arm and chemo arm who received at least 1 dose of study drug and who had an EORTC-QLQ-C30 assessment at baseline were included in the analysis. Per protocol, the pembro arm was compared to the chemo arm separately and is not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 314 | 0 | 311
Months | 8.0 [5.9 to 10.3] |  | 4.5 [2.8 to 8.2]
Statistical Analysis 1: Comparison: Pembrolizumab + ST Chemotherapy (Pembro Combo) vs ST Chemotherapy (Chemo); TTD in GHS/QoL combined score was compared between all participants of the pembro combo arm and the chemo arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Hazard Ratio (HR) = 0.78, 95% CI 2-sided [0.62 to 1.00]

19. Secondary Outcome: Pembro vs Chemo: Change From Baseline To Week 18 in the EORTC QLQ-C30 GHS/QoL Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the Global Health Status (GHS) question "How would you rate your overall health during the past week?" (Item 29) and the Quality of Life (QoL) question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Using linear transformation, raw scores were standardized so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. Per protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared between all participants of the pembro arm and the chemo arm as a pre-specified secondary analysis. As specified by the protocol, change from baseline to Week 18 in the GHS/QoL combined score was compared separately between all participants of the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Baseline, Week 18
Population: All participants in the ITT population randomized to the pembro arm and chemo arm who received at least 1 dose of study drug and who completed at least 1 EORTC-QLQ-C30 assessment were included in the analysis. Per protocol, the pembro combo arm was compared to the chemo arm separately and is not included in this analysis.
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a Scale
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 301 | 337
Score on a Scale |  | -1.89 [-5.04 to 1.26] | -0.95 [-3.95 to 2.06]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); Change from baseline to Week 18 in EORTC-QLQ-C30 GHS/QoL combined score was compared between all participants of the pembro arm and the chemo arm. Comparison based on cLDA model with GHS/QoL score as response variable, and with treatment by study visit interactions and stratification factors (investigator's choice of chemotherapy [cisplatin or carboplatin] and PD-L1 status [CPS<10 vs. CPS≥10]) at baseline as covariates; Test type: Other; No formal hypothesis testing was performed; Difference in LS Means = -0.94, 95% CI 2-sided [-5.06 to 3.18]

20. Secondary Outcome: Pembro vs Chemo: TTD in the EORTC-QLQ-C30 GHS/QoL (Items 29 and 30) Combined Score
Description: EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients. Participant responses to the GHS question "How would you rate your overall health during the past week?" (Item 29) and the QoL question "How would you rate your overall quality of life during the past week?" (Item 30) were scored on a 7-point scale (1=Very Poor to 7=Excellent). Raw scores were standardized by linear transformation so that scores ranged from 0 to 100, with a higher score indicating a better overall outcome. TTD in GHS/QoL was defined as the time from first dose date to the first onset of a ≥10 point decrease from baseline in GHS/QoL combined score without confirmation. Per protocol, TTD in GHS/QoL combined score was compared between the pembro arm and chemo arm. TTD in GHS/QoL combined score was compared separately between the pembro combo arm and chemo arm and is presented earlier in the record.
Time Frame: Baseline up to approximately 25 months
Population: All participants in the ITT population randomized to the pembro arm and chemo arm who received at least 1 dose of study drug and who had an EORTC-QLQ-C30 assessment at baseline were included in the analysis. Per protocol, the pembro combo arm was compared to the chemo arm separately and is not included in this analysis.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) | Pembrolizumab (Pembro) | ST Chemotherapy (Chemo)
Number analyzed (Participants) | 0 | 275 | 311
Months |  | 3.6 [2.1 to 5.2] | 4.5 [2.8 to 8.2]
Statistical Analysis 1: Comparison: Pembrolizumab (Pembro) vs ST Chemotherapy (Chemo); TTD in GHS/QoL combined score was compared between all participants of the pembro arm and the chemo arm. Comparison based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by investigator's choice of chemotherapy (cisplatin or carboplatin) and PD-L1 status (CPS<10 vs. CPS≥10) at baseline; Test type: Other; No formal hypothesis testing was performed; Hazard Ratio (HR) = 1.18, 95% CI 2-sided [0.93 to 1.49]

ADVERSE EVENTS:
Time Frame: Up to approximately 70 months
Description: All-Cause Mortality reported for all randomized participants by course. Serious and Other AEs include all treated participants according to treatment received. Per protocol, MedDRA preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" unrelated to drug excluded as AEs.
Groups:
- Pembrolizumab + ST Chemotherapy (Pembro Combo) First Course: Participants received pembrolizumab 200 mg IV on Day 1 of each 3-week cycle (Q3W) for a maximum of 35 doses PLUS ST chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle, OR carboplatin at an area under the curve 5 (AUC 5) (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle.
- Pembrolizumab (Pembro) First Course: Participants received pembrolizumab 200 mg intravenously (IV) on Day 1 of each 3-week cycle (Q3W) for a maximum of 35 doses.
- ST Chemotherapy (Chemo) First Course: Participants received ST chemotherapy with EITHER cisplatin 70 mg/m^2 IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine IV infusion 1,000 mg/m^2 on Day 1 and Day 8 of each 3-week cycle OR carboplatin at AUC 5 (or AUC 4.5 if required per local guidelines) IV on Day 1 (or Day 2 if required per local guidelines) of each 3-week cycle plus gemcitabine 1,000 mg/m^2 IV on Day 1 and Day 8 of each 3-week cycle.
- Pembrolizumab + ST Chemotherapy (Pembro Combo) Second Course: Eligible participants who stopped the initial course of pembrolizumab (200 mg IV Q3W for up to 35 treatments [approximately 2 years]) administered in combination with ST chemotherapy, and experienced Stable Disease (SD) or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (up to approximately 1 additional year).
- Pembrolizumab (Pembro) Second Course: Eligible participants who stopped the initial course of pembrolizumab (200 mg IV Q3W for up to 35 treatments [approximately 2 years]) with SD or better but progressed after discontinuation initiated a second course of pembrolizumab at the investigator's discretion for up to 17 cycles (up to approximately 1 additional year).
Arm/Group | Pembrolizumab + ST Chemotherapy (Pembro Combo) First Course | Pembrolizumab (Pembro) First Course | ST Chemotherapy (Chemo) First Course | Pembrolizumab + ST Chemotherapy (Pembro Combo) Second Course | Pembrolizumab (Pembro) Second Course
All-Cause Mortality (participants affected / at risk) | 283/351 | 244/307 | 300/352 | 4/14 | 8/15
Serious Adverse Events (participants affected / at risk) | 189/349 | 145/302 | 138/342 | 0/14 | 0/15
Other Adverse Events (participants affected / at risk) | 345/349 | 275/302 | 337/342 | 0/14 | 1/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + ST Chemotherapy (Pembro Combo) First Course (N=349) | Pembrolizumab (Pembro) First Course (N=302) | ST Chemotherapy (Chemo) First Course (N=342) | Pembrolizumab + ST Chemotherapy (Pembro Combo) Second Course (N=14) | Pembrolizumab (Pembro) Second Course (N=15)
Anaemia (Blood and lymphatic system disorders) | 15 (15) | 6 (8) | 19 (19) | 0 (0) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 9 (9) | 0 (0) | 11 (11) | 0 (0) | 0 (0)
Haematotoxicity (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 10 (10) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 12 (15) | 0 (0) | 10 (11) | 0 (0) | 0 (0)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure (Cardiac disorders) | 0 (0) | 5 (5) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dolichocolon (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Odontogenic cyst (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Adrenocortical insufficiency acute (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adrenocorticotropic hormone deficiency (Endocrine disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia of malignancy (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypopituitarism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thyroiditis (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epiretinal membrane (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune colitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 2 (4) | 1 (1) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 3 (4) | 5 (5) | 4 (4) | 0 (0) | 0 (0)
Enterocolitis haemorrhagic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Enterocolonic fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal fistula (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Large intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Mechanical ileus (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rectal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Short-bowel syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Subileus (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Asthenia (General disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 6 (6) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypothermia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Medical device site laceration (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 6 (7) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cirrhosis alcoholic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Liver injury (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sarcoidosis (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal infection (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute hepatitis B (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Bacterial diarrhoea (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 3 (3) | 4 (4) | 3 (3) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device related infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Device related sepsis (Infections and infestations) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterobacter bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Escherichia urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Intervertebral discitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Parotid abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic abscess (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Periodontitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peritonitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 8 (8) | 6 (7) | 6 (6) | 0 (0) | 0 (0)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 5 (5) | 6 (6) | 3 (3) | 0 (0) | 0 (0)
Pyelonephritis acute (Infections and infestations) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyonephrosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash pustular (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 3 (3) | 1 (2) | 4 (4) | 0 (0) | 0 (0)
Septic arthritis staphylococcal (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stoma site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 31 (65) | 19 (22) | 22 (28) | 0 (0) | 0 (0)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 13 (15) | 7 (7) | 7 (7) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal wound dehiscence (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural discharge (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pneumothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Urethral injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urostomy complication (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Anticoagulation drug level above therapeutic (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
International normalised ratio increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Liver function test increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 0 (0) | 7 (7) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 11 (13) | 1 (1) | 15 (24) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Diabetes mellitus (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fluid retention (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fulminant type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 5 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral venous thrombosis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 2 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Dementia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Encephalitis autoimmune (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Myoclonus (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Polyneuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device occlusion (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 17 (21) | 13 (15) | 9 (9) | 0 (0) | 0 (0)
Autoimmune nephritis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder tamponade (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 9 (10) | 14 (20) | 3 (3) | 0 (0) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prerenal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tubulointerstitial nephritis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ureteric obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urethral fistula (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 5 (5) | 1 (1) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 4 (5) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pharyngeal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 3 (3) | 4 (4) | 0 (0) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arterial haemorrhage (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 4 (4) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Embolism (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypovolaemic shock (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic venous thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Peripheral ischaemia (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vascular pain (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + ST Chemotherapy (Pembro Combo) First Course (N=349) | Pembrolizumab (Pembro) First Course (N=302) | ST Chemotherapy (Chemo) First Course (N=342) | Pembrolizumab + ST Chemotherapy (Pembro Combo) Second Course (N=14) | Pembrolizumab (Pembro) Second Course (N=15)
Anaemia (Blood and lymphatic system disorders) | 227 (334) | 75 (103) | 210 (303) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 31 (60) | 0 (0) | 25 (55) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 126 (274) | 2 (2) | 129 (281) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 86 (175) | 2 (2) | 89 (180) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 34 (43) | 30 (33) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 41 (51) | 29 (35) | 29 (31) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 12 (15) | 9 (11) | 26 (26) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 124 (155) | 56 (70) | 107 (140) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 102 (136) | 58 (81) | 73 (91) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 14 (16) | 6 (6) | 22 (27) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 19 (20) | 1 (1) | 6 (7) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 180 (279) | 43 (53) | 154 (247) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 22 (28) | 13 (14) | 18 (20) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 91 (142) | 33 (43) | 72 (108) | 0 (0) | 0 (0)
Asthenia (General disorders) | 84 (138) | 42 (50) | 84 (120) | 0 (0) | 0 (0)
Fatigue (General disorders) | 147 (199) | 78 (94) | 122 (150) | 0 (0) | 0 (0)
Malaise (General disorders) | 12 (13) | 3 (3) | 20 (23) | 0 (0) | 0 (0)
Mucosal inflammation (General disorders) | 20 (23) | 4 (4) | 9 (15) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 47 (55) | 27 (34) | 44 (48) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 77 (112) | 43 (58) | 41 (62) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 19 (27) | 14 (20) | 16 (16) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 26 (31) | 10 (14) | 10 (10) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 70 (109) | 62 (93) | 48 (55) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 54 (106) | 20 (22) | 21 (35) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 52 (93) | 21 (33) | 20 (23) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 23 (31) | 17 (19) | 11 (21) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 68 (105) | 38 (39) | 39 (51) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 77 (174) | 2 (3) | 69 (152) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 78 (159) | 5 (5) | 79 (169) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 38 (43) | 38 (39) | 22 (23) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 55 (136) | 1 (1) | 51 (109) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 121 (147) | 72 (79) | 95 (122) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 23 (54) | 14 (16) | 7 (14) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 34 (60) | 24 (36) | 17 (22) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 19 (28) | 19 (22) | 7 (8) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 33 (61) | 19 (28) | 11 (12) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 39 (53) | 9 (10) | 24 (26) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 31 (47) | 25 (36) | 16 (23) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 (70) | 35 (41) | 24 (25) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 50 (67) | 37 (43) | 19 (22) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 32 (36) | 24 (27) | 14 (17) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 45 (54) | 19 (23) | 36 (41) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 25 (28) | 8 (8) | 28 (30) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 42 (52) | 17 (23) | 27 (33) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 24 (32) | 2 (2) | 20 (23) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 35 (40) | 19 (19) | 16 (18) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 19 (22) | 9 (10) | 7 (10) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 53 (66) | 31 (33) | 18 (19) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 55 (65) | 30 (34) | 28 (30) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 55 (62) | 34 (40) | 36 (40) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 22 (25) | 3 (3) | 23 (31) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 21 (29) | 1 (1) | 14 (22) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 26 (26) | 0 (0) | 28 (29) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 12 (13) | 18 (19) | 7 (7) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 80 (109) | 66 (89) | 17 (21) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 82 (108) | 40 (57) | 24 (33) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 23 (26) | 13 (17) | 10 (10) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the Sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/05/NCT02853305/Prot_SAP_001.pdf